CLINICAL TRIAL: NCT05877118
Title: Improving Availability of Intranasal Naloxone Rescue for Opioid Overdose
Brief Title: Improving Availability of Intranasal Naloxone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Hartford HealthCare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HHC-2023-0079
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Opioid Overdose
Keywords: Naloxone; Overdose education
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard education (Active Comparator): Written instructions and information communicated to the patient through MyChart. The following four key points are covered: (1) When someone overdoses on opiates, their breathing will get very slow and may stop (2) Naloxone is a safe life-saving medication that can reverse an opioid overdose (3) You give someone naloxone by injecting it through the nostril, (4) If a first dose of naloxone does not work after about 3 minutes, give a second dose.
  Interventions: Behavioral: Standard education
- Enhanced Overdose Education (EOE) (Experimental): A one-page education pamphlet handed to participants and their identified support individual and a 4-minute video clip that will be viewed in the hospital and emailed or texted to both. EOE is purposefully brief and intended to increase uptake by participants and their support network who may not be motivated or willing to engage in face-to-face or extensive education. The pamphlet and video both emphasize the Why and How. That is, the significance of naloxone in decreasing the likelihood of death following an overdose while providing simple instructions on how to use the nasal kit. They also emphasize an important point missing in standard education: to tell others in the support network where it is and how to use it.
  Interventions: Behavioral: Enhanced Overdose Education (EOE)

INTERVENTIONS:
Behavioral: Enhanced Overdose Education (EOE) — EOE was adapted by Co-I Dr. Monique Miley at HHC's premier addiction hospital-The Rushford Center. It follows the guidelines set by Co-PI Jonathan Craig Allen when working with opioid patients reluctant to obtain naloxone:
  * Express confidence in naloxone
  * Provide a clear statement about suitability (You are an excellent candidate for naloxone)
  * Begin discussion using presumptive language (You must be ready for an overdose)
  Arms: Enhanced Overdose Education (EOE)
Behavioral: Standard education — Written instructions that accompany a kit prescription in many EDs throughout the country.
  Arms: Standard education

SUMMARY:
While there is a lifesaving medication called naloxone that can reverse the deadly effects of opioid overdose, patients often fail to fill the prescription at the pharmacy when it is prescribed. This is particularly concerning and true in those at the highest risk of death-those who end up in the emergency department for opioid overdose. The goal of this study is to compare the impact of different overdose education on naloxone prescription fill rates in opioid users being discharged from our hospital emergency department. You will receive either (a) written education about naloxone through their MyChart account, or (b) a concise one-page handout and 4-minute video clip reviewed with the participant and a support individual (family/friend) prior to discharge.

DETAILED DESCRIPTION:
The rates of opioid overdose and overdose deaths in Connecticut have increased dramatically in the past decade. While there is a lifesaving medication called naloxone that can reverse the deadly effects of opioid overdose, patients often fail to fill the prescription at the pharmacy when it is prescribed. This is particularly concerning and true in those at the highest risk of death-those who end up in the emergency department for opioid overdose. Indeed, a recent national study by the University of Michigan found that from 2001 to 2016 less than 1% of patients filled their prescription for naloxone following ED discharge. To address this problem, The investigators propose a prospective randomized clinical trial comparing an experimental education intervention that may improve prescription fill rate against the current standard of care at the Hartford Hospital ED (HH-ED). Our primary aim is to provide preliminary data on the impact of an enhanced overdose education (EOE) delivered at the HH-ED, on intranasal naloxone rescue kit prescription fill rates in opioid users. The investigators hypothesize that compared to those who receive standard education (written instructions, current standard of care), opioid users who receive EOE while being discharged from the emergency department will be more likely to fill the prescription for an intranasal naloxone rescue kit within one month of hospital discharge. Our secondary aim is to obtain preliminary data on the impact of EOE, delivered at the HH-ED, on naloxone rescue kit knowledge. The investigators hypothesize that compared to the current standard education, opioid users and their support network, who receive EOE while being discharged from the emergency department, will retain more educational content about naloxone rescue kits at one-month post ED visit. In exploratory fashion, the investigators will also qualitatively examine reasons the kit was or was not filled. The long-term, overarching goal of this line of research is to reduce mortality in opioid users, starting with increasing the likelihood that rescue kit prescriptions will be filled.

ELIGIBILITY:
Inclusion Criteria:

-Patients will be in the process of being discharged from Hartford Hospital ED with a naloxone kit prescription following opiate or opioid intoxication/poisoning, use of illicit opioids or prescription opioids, or opioid injection use-related conditions

Exclusion Criteria:

* Patient has previously received the standard naloxone kit education or has a known allergy to naloxone and/or kit constituents
* Patient or support network does not speak English
* Patient is in police custody
* Patient is not being discharged home from the ED.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prescription fill rate | 1 month
  Pharmacy records/survey to determine if naloxone kit prescription was filled

SECONDARY OUTCOMES:
Education content survey | 1 month
  Questionnaire measuring how much of education was retained and reasons for filling or not filling prescription

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Allen, MD, Principal Investigator — Hartford HealthCare
Locations (2):
- United States (2):
  - Hartford Hospital Emergency Department, Hartford, Connecticut
  - Olin Neuropsychiatry Research Center, Hartford, Connecticut

IPD SHARING:
Plan to Share IPD: No